CLINICAL TRIAL: NCT03185234
Title: Therapeutischer Einsatz Der Schwachen Gleichstromstimulation (tDCS) Bei Motorisch-kognitiven Defiziten Nach Schlaganfall
Brief Title: Rehabilitating (Stroke-induced) Apraxia With Direct Current Stimulation
Acronym: RAdiCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Gereon R. Fink, Univ.-Prof. Dr. med., University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Uni-Koeln-3033; U1111-1195-2536 (Other: WHO); DRKS00012292 (Registry Identifier: DRKS)
Record Dates: First submitted 2017-05-31; First posted 2017-06-14 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Stroke; Apraxia
Keywords: tDCS
MeSH Terms: conditions — Stroke; Apraxias | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS (Active Comparator): Anodal tDCS at an intensity of 2 mA is applied for 10 minutes at a time on 5 consecutive days. The anodal electrode is placed over the left parietal cortex (P3 in 10/20 EEG) of the lesioned hemisphere, the cathodal electrode is located supraorbital on the right side. Motor tasks are performed before and after the stimulation.
  Interventions: Device: anodal tDCS
- Sham tDCS (Sham Comparator): Sham stimulation is applied for 10 minutes at a time on 5 consecutive days. One electrode is placed over the left parietal cortex (P3 in 10/20 EEG) of the lesioned hemisphere and a second electrode supraorbital on the right side. Motor tasks are performed before and after the stimulation.
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: anodal tDCS — 2 mA, 10 min, 5 sessions
  Other Names: neuroConn DCS, model no. 008
  Arms: Real tDCS
Device: sham tDCS — sham stimulation, 10 min, 5 sessions
  Other Names: neuroConn DCS, model no. 008
  Arms: Sham tDCS

SUMMARY:
The objective of the clinical trial is to investigate whether weak transcranial direct current stimulation (tDCS) can ameliorate the motor cognitive deficit apraxia during stroke rehabilitation. Stroke patients with apraxia will either receive a real stimulation or a sham stimulation (placebo) for 10 minutes at a time on 5 consecutive days during their in-patient stay in a rehabilitation center. Additionally, motor tasks are performed before and after the stimulation. The effect of the weak current stimulation on motor function is assessed 3-4 days after the last stimulation and 3 months after enrollment.

DETAILED DESCRIPTION:
Despite the high incidence of the motor cognitive deficit apraxia after left-hemispheric stroke, evidence-based therapies do not exist. This randomized controlled clinical trial (RCT) investigates whether anodal transcranial direct current stimulation (tDCS) as an add-on therapy during neuro-rehabilitation can ameliorate apraxic deficits in patients with left hemisphere stroke. Therefore, anodal tDCS is applied over the parietal cortex of the left, lesioned hemisphere with an intensity of 2 mA for 10 minutes at a time on 5 consecutive days in combination with motor tasks before and after the stimulation. The effect of the stimulation is compared to a sham stimulation. Moreover, application of a pre-programmed study mode ensures a double-blind study design (patient and investigator). The performance in the apraxia test KAS (Cologne Apraxia Screening) 3-4 days after the last stimulation, compared to baseline, serves as primary endpoint of the study. Secondary endpoints are evaluated using various apraxia tests, motor tests and neuropsychological tests 3-4 days after the last stimulation and 3 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* left hemispheric ischemic stroke in the subacute/ chronic phase (>10 days and <180 days post-stroke)
* clinical confirmation of apraxia by KAS (Cologne Apraxia Screening), Cut-off ≤ 76/ 80 points;
* age 18 - 90 years;
* written Informed Consent

Exclusion Criteria:

* pregnancy, breastfeeding and women without exclusion of pregnancy
* patients with clinical manifestation of a stroke prior to the index-stroke
* malignant disease with affection of central nervous system
* life expectancy <12 months
* current addiction to alcohol or drugs or other addictive disease (exception: nicotine)
* current clinically manifest psychiatric disorders, such as schizophrenia or severe depressive episode
* epileptic seizure within the past two years
* continuous medication during the intervention phase with benzodiazepine, antipsychotics of high potential and anti-epileptic drugs taken for prophylaxis of epileptic seizures
* enrollment in other studies with brain stimulation in the time period after the index stroke
* heart pacemaker
* electrodes for deep brain stimulation or other metal implants in the head (expected are dental fillings and inlays)
* craniectomy or trepanation
* vulnerable skin lesions at electrode positions
* poor motivation/ cooperation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
KAS (Cologne Apraxia Screening) | 3-4 days after stimulation
  Degree of apraxia

SECONDARY OUTCOMES:
KAS (Cologne Apraxia Screening) | 3 months after enrollment
  Degree of apraxia
Goldenberg Imitation | 3-4 days after stimulation, and 3 months after enrollment
  Degree of apraxia
de Renzi Imitation | 3-4 days after stimulation, and 3 months after enrollment
  Degree of apraxia
de Renzi actual tool use | 3-4 days after stimulation, and 3 months after enrollment
  Degree of apraxia
Action Research Arm Test (ARAT) | 3-4 days after stimulation, and 3 months after enrollment
  Motor function
Jebsen Taylor Hand Function Test (JTHFT) | 3-4 days after stimulation, and 3 months after enrollment
  Motor function
Gripforce (Vigorimeter) | 3-4 days after stimulation, and 3 months after enrollment
  Motor function
Strength of hands (MRC) | 3-4 days after stimulation, and 3 months after enrollment
  Motor function
National Institute of Health Stroke Scale (NIHSS) | enrollment
  Impairment by stroke
modified Ranking Scale (mRS) | 3-4 days after stimulation, and 3 months after enrollment
  Impairment by stroke
Aphasia Check List (ACL-K) | 3-4 days after stimulation, and 3 months after enrollment
  Aphasia

CONTACTS AND LOCATIONS:
Overall Officials: Gereon R. Fink, Univ-Prof., Principal Investigator — University Hospital Cologne
Locations (2):
- Germany (2):
  - Rehabilitationszentrum Godeshöhe e.V., Bonn, North Rhine-Westphalia
  - MediClin Fachklinik Rhein/Ruhr für Neurologie, Essen, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kleineberg NN, Richter MK, Becker I, Weiss PH, Fink GR. Verum versus sham tDCS in the treatment of stroke-induced apraxia: study protocol of the randomized controlled trial RAdiCS -"Rehabilitating (stroke-induced) Apraxia with direct Current Stimulation". Neurol Res Pract. 2020 Mar 4;2:7. doi: 10.1186/s42466-020-0052-y. eCollection 2020. PMID 33324913